CLINICAL TRIAL: NCT03641599
Title: Assessment Right Ventricular Systolic Function in Heart Failure With Preserved, Reduced and Mid-range Ejection Fraction
Brief Title: Right Ventricular Function in Heart Failure
Status: Completed | Type: Observational
Sponsor: shaimaa Mostafa (Other)
Responsible Party: Sponsor-Investigator, shaimaa Mostafa, assistant professor of cardiovascular medicicne, Benha University
Organization: Benha University (Other)
Other Study IDs: RV
Record Dates: First submitted 2018-08-17; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Assessment of the RV Function in Patients With Heart Faliure
Keywords: RV systolic function; HFpEF; HFmrEF; HFrEF
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- heart failure with preserved ejection fraction
  Interventions: Diagnostic Test: echocardiography
- heart failure with mid range ejection fraction
  Interventions: Diagnostic Test: echocardiography
- heart failure with reduced ejection fraction
  Interventions: Diagnostic Test: echocardiography

INTERVENTIONS:
Diagnostic Test: echocardiography — echocardiographic assessment of the RV and LV systolic function

SUMMARY:
Only a few studies evaluated the RV systolic function in the three categories of HF, regarding the importance of understanding changes in RV function on clinical presentation and outcome; it was essential to understand the prevalence and severity of RV dysfunction among the three groups and the degree of correlation between RV with LV systolic function.

ELIGIBILITY:
Inclusion Criteria:

-

Adult patients of both gender who have the followiong criteria :

(i) symptoms with or without signs of HF (ii) elevated natriuretic peptides (BNP ≥35pg/ mL or NT-proBNP≥125pg/mL) (iii) relevant structural heart disease: left ventricle hypertrophy (left ventricular mass index ≥115 g/m2 for males and ≥95 g/m2 for females) or left atrial enlargement (>34 mL/m2) or diastolic dysfunction (E/e'≥13 and a mean e' septal and lateral wall <9 cm/s) were included.

Then patients were classified according to EF into HFpEF>50%, HFrEF<40% and HFmrEF >40% and <50%

Exclusion Criteria:

Patients with chronic obstructive pulmonary disease history of pulmonary embolism patients with respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HFpEF>50%, HFrEF<40% and HFmrEF >40% and <50%
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
assessment of the RV systolic dysfunction in patients with heart failure | 1.5 year
  degree and prevalence of the RV systolic dysfunction in patients with heart failure with preserved, mid-range and decreased ejection fraction

REFERENCES:
- [Derived] Mostafa S. Assessment of right ventricular systolic function in heart failure with preserved, reduced and mid-range ejection fraction. Indian Heart J. 2019 Sep-Oct;71(5):406-411. doi: 10.1016/j.ihj.2019.11.252. Epub 2019 Nov 20. PMID 32035524